CLINICAL TRIAL: NCT03951974
Title: A Social Emotion Regulation Intervention in MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PC 8-19
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis; Emotional Disturbances
Keywords: emotion regulation; social regulation of emotion
MeSH Terms: conditions — Multiple Sclerosis; Affective Symptoms; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants in the experimental group will receive training in utilizing social regulation of emotion strategies in an individualized format. They will meet with an interventionist for 5 weeks (1 in-person session and 4 telephone sessions) for 1-1.5 hours each week, and keep a journal documenting their emotion challenges and regulation strategy use.
  Interventions: Behavioral: Social Emotion Regulation Strategy Development
- Control (Other): Participants in the control group will not receive training in utilizing social regulation of emotion strategies. While they will still meet with the interventionist on the same schedule and for approximately the same length of time, they will simply be asked to report the emotion regulation strategies that they naturally employ. They will also keep a journal documenting their emotion challenges and regulation strategy use.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Social Emotion Regulation Strategy Development — Participants will work one-on-one with an interventionist to develop goals (in the form of implementation intentions) to develop social emotion regulation strategies to combat frequent emotional challenges.
  Arms: Experimental
Behavioral: Control — Participants will work one-on-one with an interventionist to report on their frequent emotional challenges, and report the emotion regulation strategies that they frequently use to combat them.
  Arms: Control

SUMMARY:
The current project will examine effectiveness of an intervention based on the concept of the social regulation of emotion. The intervention is designed to improve well-being in individuals with MS by leveraging participants' existing social support. Effectiveness will be tested on a sample of 42 individuals with MS, half of whom will receive the intervention and half of which will receive an inactive control. Investigators will document changes resulting from treatment on self-reported levels of stress, depression, and quality of life. Intervention evaluation will expand scientific knowledge of emotion regulation disruption in MS, and potentially identify a novel and highly efficient means of treatment.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a progressive and debilitating neurological disease which not only affects a patient's physical health, but also adversely affects their mental health. Depressed mood is common in MS, and poor mental health in individuals with MS has wide-ranging consequences on social relationships and community integration. The preponderance of negative emotions and sparsity of positive emotions in MS are attributable in part to ineffective emotion regulation strategies. Thus, the clinical trial seeks to evaluate the effectiveness of an intervention which instructs individuals on using the social regulation of emotion.

The social regulation of emotion occurs when a one's emotional state benefits from an interaction with another person, such as when seeking comfort from a trusted friend. The current intervention was designed to leverage existing social relationships for emotional support in a manner which should strengthen the perception of social support and also reinforce existing relationships. The primary goal of this trial is to examine changes in mental well-being after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis diagnosis
* English language fluency

Exclusion Criteria:

* currently taking steroids or benzodiazepines
* within 30 days of an exacerbation
* history of substance abuse
* diagnosis of bipolar, schizophrenia, epilepsy, stroke

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2021-07-09 (Estimated); Study Completion 2021-07-09 (Estimated)

PRIMARY OUTCOMES:
Well-being: Depression | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 6)
  Change in scores on a self-report questionnaire of depression (the Center for Epidemiologic Studies Depression Scale, a 20-item scale with higher scores indicating greater depression)
Well-being: Stress | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 6)
  Change in scores on a self-report questionnaire of stress (the Perceived Stress Scale, a 10-item scale with higher scores reflecting higher stress)
Well-being: Quality of life | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 6)
  Change in scores on a self-report questionnaire of quality of life (the Satisfaction with Life Scale, a five item scale where higher scores reflect higher satisfaction)

SECONDARY OUTCOMES:
Perceived social support | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 6)
  Change in scores on a self-report questionnaire of perceived social support (the Multidimensional Scale of Perceived Social Support, a 12-item scale where higher scores reflect greater support)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Lancaster, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Individual participant data that underlie publication in an article will be shared.
Time Frame: Immediately following publication. No end date.
Access Criteria: Any purpose